CLINICAL TRIAL: NCT03077594
Title: Prospective Characterization of the Neo-squamous Epithelial Barrier Following Successful Endoscopic Therapy in Barrett's Esophagus
Brief Title: Characterization of the Neo-squamous Epithelial Barrier
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Other Study IDs: 16-005490
Record Dates: First submitted 2017-02-01; First posted 2017-03-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Barrett's Esophagus With Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Esophageal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successfully ablated patients: Mucosal impedance will be performed at the time of clinically indicated endoscopy. Research biopsies will be obtained during clinically indicated endoscopy.
  Interventions: Device: Mucosal Impedance; Other: Research Biopsies
- Successfully ablated patients - VLE: Mucosal impedance will be performed at the time of clinically indicated endoscopy. Research biopsies will be obtained during clinically indicated endoscopy. Volumetric laser endomicroscopy (VLE) will be done.
  Interventions: Device: Mucosal Impedance; Other: Research Biopsies; Device: Volumetric Laser Endomicroscopy

INTERVENTIONS:
Device: Mucosal Impedance — Aim 1: Mucosal impedance will be measured by an endoscopic probe 1 cm above the gastroesophageal junction, 5 cm above the gastroesophageal junction and in the proximal esophagus in an area not exposed to the index therapeutic radiofrequency ablation. Aim 2: Mucosal impedance will be measured 1 cm above gastroesophageal junction, 1 cm below previous squamous columnar junction, 1 cm above previous squamocolumnar junction.
Other: Research Biopsies — Aim 1: Research biopsies will be obtained at 1 cm above the gastroesophageal junction, 5 cm above the gastroesophageal junction, and in the proximal esophagus in an area not exposed to the index therapeutic radiofrequency ablation. Aim 2: Aim 2: Research biopsies will be taken 1 cm above gastroesophageal junction, 1 cm below previous squamous columnar junction, 1 cm above previous squamocolumnar junction.
Device: Volumetric Laser Endomicroscopy — Aim 2: Volumetric laser endomicroscopy will be done and marked at 1 cm above gastroesophageal junction, 1 cm below previous squamous columnar junction, 1 cm above previous squamocolumnar junction.
  Groups: Successfully ablated patients - VLE

SUMMARY:
To prospectively assess the functional aspects of the the esophageal squamous epithelial barrier and correlate this with tissue inflammation and intercellular space dilation in patients who have successfully completed endoscopic radiofrequency ablation versus balloon cryotherapy for Barrett's Esophagus related metaplasia.

DETAILED DESCRIPTION:
The investigators will measure and correlate mucosal impedance (measured using a novel endoscopic mucosal impedance catheter), intercellular space as measured with transmission electron microscopy and tissue levels of prostaglandin E2 in patients undergoing surveillance following successful endoscopic therapy (defined as two negative endoscopic surveillance histology for intestinal metaplasia).

Mucosal impedance will be measured by an endoscopic probe. Research biopsies will also be obtained for measurement of tissue levels of prostaglandin E2 and intracellular space with transmission electron microscopy.

Volumetric laser endomicroscopy will measure the precise thickness of and area of subsquamous structures underneath the neosquamous epithelium.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-90) who underwent an ablative program for BE

Exclusion Criteria:

* Patients that have not achieved complete remission of intestinal metaplasia.
* Patients unable to consent.
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have successfully completed endoscopic ablation (one endoscopy with no evidence of intestinal metaplasia).
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Mucosal Impedance as measured by an endoscopic probe | Up to two years
  Assess the mucosal impedance of neosquamous epithelium after successful treatment of Barrett's Esophagus.

SECONDARY OUTCOMES:
Tissue levels of prostaglandin E2 | Up to two years
  Assess the levels of prostaglandin E2 in neosquamous epithelium after successful treatment of Barrett's Esophagus.
Intracellular space | Up to two years
  Assess the intercellular space in neosquamous epithelium following successful treatment of Barrett's Esophagus with use of transmission electron microscopy.
Volumetric Laser Endomicroscopy | Up to two years
  Assess and measure precise thickness of and area of subsquamous structions underneath the neosquamous epithelium.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Iyer, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials